CLINICAL TRIAL: NCT02928601
Title: Does Prophylactic Ondansetron Reduce Norepinephrine Consumption in Patients Undergoing Caesarean Section With Spinal Anesthesia?
Brief Title: Norepinephrine Consumption After Prophylactic Ondansetron
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Feride Karacaer, Specialist doctor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NAOS1
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Maternal Hypotension
MeSH Terms: interventions — Ondansetron; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron (Experimental)
  Interventions: Drug: Ondansetron
- Saline (Active Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ondansetron — After spinal anesthesia, half of the patients will be given intravenous 8 mg ondansetron.
  Arms: Ondansetron
Drug: Saline — After spinal anesthesia, half of the patients will be given intravenous 2 mlt saline.
  Arms: Saline

SUMMARY:
This study evaluates the effect of prophylactic ondansetron on the incidence of spinal hypotension and vasopressor consumption in caesarean section patients using norepinephrine treatment. Half of participants receive ondansetron before spinal anesthesia while the other half receive saline.

DETAILED DESCRIPTION:
Spinal hypotension in cesarean section patients can occur vigorously and may lead to cardiovascular collapse. If doesn't treated precipitously, It can cause maternal hypotension, nausea and vomiting and fetal acidosis. Recently norepinephrine has been proposed for the prevention and treatment of spinal hypotension with less tendency to decrease HR and CO. It has been reported that ondansetron can be used for prophylaxis and treatment of nausea and vomiting, may also reduce the vasopressor requirement in patients undergoing caesarean section with spinal anesthesia. The aim of the present study is to assess the effect of prophylactic ondansetron on norepinephrine consumption and incidence of spinal hypotension, and side effects such as maternal nausea, vomiting and bradycardia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II patients
* Between the ages of 18 and 40 years
* Scheduled for elective caesarean section with spinal anesthesia

Exclusion Criteria:

* History of hypertension
* History of severe hepato-renal disease,
* sensitivity or contraindication to ondansetron,
* Drug or alcohol abuse
* Contraindication to regional anesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Norepinephrine consumption | During the cesarean operation
  Whenever systolic arteriel pressure falls below 100 mmHg or below 20% of the preoperative baseline value in both groups norepinephrine (5 µg) will be administered intravenously and total consumption will be recorded.

SECONDARY OUTCOMES:
Bradicardia | During the cesarean operation
  Heart rate lower than 60 beat /min will be treated with iv 0.5 mg of atropine and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hakkı Ünlügenç, Professor, Study Director — Cukurova University
Locations (1):
- Çukurova University, Adana, Turkey (Türkiye)

REFERENCES:
- [Result] Gao L, Zheng G, Han J, Wang Y, Zheng J. Effects of prophylactic ondansetron on spinal anesthesia-induced hypotension: a meta-analysis. Int J Obstet Anesth. 2015 Nov;24(4):335-43. doi: 10.1016/j.ijoa.2015.08.012. Epub 2015 Aug 22. PMID 26421701
- [Result] Wang Q, Zhuo L, Shen MK, Yu YY, Yu JJ, Wang M. Ondansetron preloading with crystalloid infusion reduces maternal hypotension during cesarean delivery. Am J Perinatol. 2014 Nov;31(10):913-22. doi: 10.1055/s-0033-1364189. Epub 2014 Feb 10. PMID 24515619